CLINICAL TRIAL: NCT05026177
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, 76-week Study Evaluating the Safety and Efficacy of Two Doses of Simufilam in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Simufilam 50 mg or 100 mg for Mild-to-Moderate Alzheimer's Disease
Acronym: REFOCUS-ALZ
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cassava Sciences, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-125-06
Record Dates: First submitted 2021-08-09; First posted 2021-08-30 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized treatments will be assigned by subject numbers in a randomly generated numeric sequence. Randomization (1:1:1) will be stratified by low or high Mini-Mental State Exam (MMSE; 16-20 and 21-27).
  The randomization code will not be revealed to study subjects, Investigators, clinical staff, study monitors or the Sponsor until all subjects have completed therapy and the database has been finalized and locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo, supplied by Cassava as coated tablets, and taken twice daily (b.i.d.) for 76 weeks
  Interventions: Drug: Placebo
- Simufilam 50 mg (Experimental): Simufilam 50 mg, supplied by Cassava as coated tablets, and taken b.i.d. for 76 weeks
  Interventions: Drug: Simufilam
- Simufilam 100 mg (Experimental): Simufilam 100 mg, supplied by Cassava as coated tablets, and taken b.i.d. for 76 weeks
  Interventions: Drug: Simufilam

INTERVENTIONS:
Drug: Simufilam — Simufilam is a novel drug candidate designed to treat and slow the progression of AD. Simufilam binds with femtomolar affinity to an altered conformation of filamin A that is present in the brain of patients with AD and critical to the toxicity of Aβ42. In this study, simufilam will be given b.i.d. for 76 weeks at a dose of 50 mg or 100 mg.
  Other Names: PTI-125
  Arms: Simufilam 100 mg; Simufilam 50 mg
Drug: Placebo — Matching placebo given b.i.d. for 76 weeks
  Arms: Placebo

SUMMARY:
A 76-week safety and efficacy study of simufilam (PTI-125) given twice daily to participants with mild-to-moderate Alzheimer's disease (AD) for 76 weeks. Approximately 1083 participants will be randomized (1:1:1) to receive either placebo, 50 mg tablets of simufilam, or 100 mg tablets of simufilam, twice daily, for 76 weeks. Clinic visits will occur 4 weeks after the baseline visit, and then every 12 weeks until the end of the study. The safety of simufilam, and its efficacy in enhancing cognition and slowing cognitive and functional decline will be evaluated.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the safety and efficacy of simufilam (PTI-125) in enhancing cognition and slowing cognitive and functional decline following 76-week, repeat-dose oral administration in participants with mild-to-moderate AD. Secondary objectives are to assess neuropsychiatric symptoms and to replicate the cerebrospinal fluid (CSF) biomarker effects observed in the two Phase 2 studies (PTI-125-03 and PTI-125-02) after 76 weeks of simufilam treatment. A third objective is to investigate the effect of simufilam treatment on plasma biomarkers as well as anatomical correlates of disease progression (brain volume [hippocampus, ventricles and whole brain]; and amyloid and tau deposition in the brain). A limited number of research sites will be invited to participate in sub-studies to assess the impact of simufilam on anatomical and biomarker endpoints, including: change from Baseline in CSF biomarkers (30 subjects/group); brain volume via magnetic resonance imaging (MRI) (50 subjects/group); and amyloid and tau positron emission tomography (PET) (40 and 50 subjects/group, respectively). Participants in both PET sub-studies will be required to have an MRI during the Screening Period and provide plasma for a biomarker sub-study. Participants in the tau PET sub-study will also provide additional plasma for a pharmacokinetic (PK) exposure response analysis. Changes from baseline for these imaging and fluid biomarkers represent additional secondary endpoints. The 90 subjects (30 per group) in the CSF sub-study will undergo lumbar puncture during the Screening Period and again at the Week 76 End-of-Treatment Visit to collect CSF biomarkers.

Safety will be evaluated by adverse event monitoring, vital signs, clinical labs, and the Columbia Suicide Severity Rating Scale at every visit. Subjects will undergo MRI during screening to ensure entry criteria are met (unless recent MRI confirms entry criteria); however, 150 subjects (50 subjects per treatment group) will also undergo repeat MRI assessments at Weeks 40 and 76 to assess both long-term safety and drug impact on brain volume as noted above. Resting electrocardiograms will be conducted at Baseline (Study Day 1) and Weeks 4, 40 and 76. A complete physical and neurological examination will be performed at screening, and brief examinations will be performed at all other visits. Weight will be measured during the Screening Period, at Baseline (Study Day 1) and at all other visits.

An independent Data Safety Monitoring Board (DSMB) will meet periodically to review subject safety assessments and determine if dosing may continue. A charter will be developed with specific guidance for the DSMB.

ELIGIBILITY:
Key Inclusion Criteria:

1. Meets National Institute on Aging and Alzheimer's Association Research Framework criteria for individuals in clinical Stage 4 or 5 of the Alzheimer's continuum.
2. Evidence for AD pathophysiology, confirmed prior to or during screening.
3. MMSE score ≥ 16 and ≤ 27 at screening.
4. Clinical Dementia Rating - Global Score must be 0.5, 1 or 2.
5. If receiving background AD medications, the dosing regimen must be stable for at least 12 weeks prior to randomization. Chronic medications for conditions other than AD (such as depression) must be prescribed at a stable dose for at least 4 weeks prior to screening.
6. The subject has not been a cigarette smoker or chewed tobacco for at least 3 years.
7. Availability of a study partner.
8. Individuals who have participated in a clinical study with an investigational drug targeting the underlying AD process may be permitted to participate in this study.
9. Completed a COVID-19 vaccine primary series ("fully vaccinated") at least 2 weeks prior to randomization or had an unambiguous COVID-19 infection diagnosed more than 3 months before the start of the Screening Period.

Key Exclusion Criteria:

1. A neurologic condition other than AD that significantly contributes to the subject's dementia.
2. Any current primary psychiatric diagnosis other than AD if it is likely to confound cognitive assessment or ability to comply with study procedures.
3. Geriatric Depression Scale (15-item) score > 8 (Note - a subject with a score > 8 may continue in screening if, in the judgment of the Investigator, the elevated score is not attributed to a major depressive episode).
4. Suicidal ideation during the past 3 months or suicidal behavior during the past 12 months.
5. Alcohol or substance use disorder within 2 years of screening.
6. MRI presence of cerebral vascular or other significant pathology.
7. History of transient ischemic attack or stroke within 12 months of screening.
8. Seizure within 12 months of screening.
9. Severe head trauma or head trauma considered likely to be contributing to the subject's cognitive impairment.
10. Sleep apnea that is considered likely to be contributing to the subject's cognitive impairment.
11. Insufficiently controlled diabetes mellitus or hypertension.
12. Body mass index < 18.5 or > 37.5.
13. History or diagnosis of clinically significant cardiac disease.
14. Currently or previously prescribed/administered aducanumab, lecanemab, or any anti-amyloid monoclonal antibody, more than 2 doses.

Ages: 50 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1125 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kupiec, MD, Study Chair — Cassava Sciences
Locations (89):
- United States (65):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Arizona Neuroscience Research, LLC, Phoenix, Arizona
  - Clinical Endpoints, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Banner Alzheimer's Institute - Tucson, Tucson, Arizona
  - North County Neurology Associates, Carlsbad, California
  - Neuro-Pain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Healthy Brain Clinic, Long Beach, California
  - California Research Insitute, Los Angeles, California
  - Shankle Clinic and Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Pacific Research Network, LLC, San Diego, California
  - Nuvance Health Medical Practice CT, Inc. - Associated Neurologists, PC, Danbury, Connecticut
  - Ki Health Partners, LLC, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Clinical Research of Brandon, LLC, Brandon, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Brain Matters Research Inc, Delray Beach, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Alphab Global Research, Jupiter, Florida
  - K2 Medical Research, Maitland, Florida
  - Mind Institute at Miami Jewish Health, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - Health Synergy Clinical Research, Okeechobee, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Intercoastal Medical Group - Sarasota, Sarasota, Florida
  - Alzheimer's Research & Treatment Center, Stuart, Florida
  - Brain Matters Research Inc, Stuart, Florida
  - USF Health - Byrd Alzheimer's Center and Research Institute, Tampa, Florida
  - Alzheimer's Research & Treatment Center, Wellington, Florida
  - Conquest Research, Winter Park, Florida
  - Columbus Memory Center, PC, Columbus, Georgia
  - Accel Research Sites - NeuroStudies, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Advocate Aurora Health, Park Ridge, Illinois
  - University of Kentucky Sanders-Brown Center on Aging, Lexington, Kentucky
  - Neurology Center of New England, Foxborough, Massachusetts
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Office of Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - MedVadis Research, Waltham, Massachusetts
  - Patient First MD, Middletown, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - The Cognitive and Research Center of New Jersey (CRCNJ), Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Albany Medical Center, Albany, New York
  - Neurological Associates of Albany, Albany, New York
  - Integrative Clinical Trials, Brooklyn, New York
  - SPRI Clinical Trials Brooklyn, Brooklyn, New York
  - Velocity Clinical Research, Formerly Clarity Clinical Research, East Syracuse, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Accellacare Research of Winston-Salem, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Neurology Diagnostics, Dayton, Ohio
  - Neuro-Behavioral Clinical Research (NBCR), North Canton, Ohio
  - Center for Cognitive Health - Portland, Portland, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Keystone Clinical Studies, LLC, Plymouth Meeting, Pennsylvania
  - KCA Neurology, PLLC, Franklin, Tennessee
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Cedar Health Research, Irving, Texas
  - The Memory Clinic - Bennington, Bennington, Vermont
  - Northwest Clinical Research Center, Bellevue, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (11):
  - OCT Research ULC DBA Okanagan Clinical Trials, Kelowna, British Columbia
  - Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia
  - Centre Hospitalier Universitaire Dr-Georges-L.-Dumont (CHUDGLD), Moncton, New Brunswick
  - True North Clinical Research - Halifax, Halifax, Nova Scotia
  - True North Clinical Research - New Minas, New Minas, Nova Scotia
  - St. Joseph's Health Care London, London, Ontario
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Recherches Neuro-Hippocampe Inc., Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
- Puerto Rico (4):
  - Santa Cruz Behavioral PSC, Bayamón
  - Inspira Clinical Research, San Juan
  - Barbara Diaz Hernandez Md Research, Inc., San Juan
  - Instituto De Neurologia Dra. Ivonne Fraga, San Juan
- South Korea (9):
  - Chonnam National University Hospital, Gwangju, Dong-gu
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Hospital, Namdong-gu, Incheon
  - Inha University Medical Center, Incheon, Jung-go
  - Kyungpook National University Chilgok Hospital, Daegu, North Gyeongsang Province
  - Korea University Anam Hospital, Seongbuk-gu, Seoul
  - HanYang University Hospital, Seongdong-gu, Seoul
  - Asan Medical Center, Seoul, Songpa-gu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kupiec JW, Porsteinsson AP, Turner RS, Hendrix S, Mallinckrodt C, Khan A, Cohen I, Liss J, Clarnette R, Park KH, Hernandez AM, Burns LH. Phase 3 randomized clinical trials of simufilam in mild-to-moderate Alzheimer's disease. J Prev Alzheimers Dis. 2026 Jan 1:100469. doi: 10.1016/j.tjpad.2025.100469. Online ahead of print. PMID 41500915

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participation in the study required each subject to have a study partner who also consented to participate for the duration of the subject's participation. Study partners were not considered independent participants. The enrollment number and number of participants detailed below represents the number of subject/study partner dyads.
Period: Overall Study
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Started | 376 (376 dyads (i.e., 376 subjects and their 376 study partners) were randomly allocated to the intervention group.) | 374 (374 dyads (i.e., 374 subjects and their 374 study partners) were randomly allocated to the intervention group.) | 375 (375 dyads (i.e., 375 subjects and their 375 study partners) were randomly allocated to the intervention group.)
Modified Intent-to-treat Population (All randomized subjects with baseline plasma P-tau181 ≥44 pg/mL or other evidence of amyloid pathology, e.g., amyloid PET) | 299 | 311 | 308
Safety Population (All subjects who received at least 1 dose of study drug) | 376 | 374 | 373
MRI Imaging Substudy Population (Subjects who consented to take part in the MRI imaging substudy and for whom there was at least one non-missing post baseline MRI assessment available) | 76 | 66 | 72
Amyloid PET Imaging Substudy Population (Subjects who consented to take part in the amyloid PET imaging substudy) | 43 | 28 | 35
Tau PET Imaging Substudy Population (Subjects who consented to take part in the tau PET imaging substudy) | 98 | 65 | 96
Plasma Biomarker Analysis Substudy Population (Subjects who consented to take part in the plasma biomarker analysis substudy) | 98 | 65 | 96
CSF Biomarker Analysis Substudy Population (Subjects who consented to take part in the CSF biomarker analysis substudy) | 51 | 45 | 43
Completed | 201 (201 dyads in the intervention group completed the study.) | 203 (203 dyads in the intervention group completed the study.) | 217 (217 dyads in the intervention group completed the study.)
Not Completed | 175 | 171 | 158
Not completed — Adverse Event | 33 | 33 | 17
Not completed — Lost to Follow-up | 7 | 6 | 8
Not completed — Noncompliance with study drug | 6 | 2 | 1
Not completed — Physician Decision | 4 | 1 | 0
Not completed — Sponsor requests subject to be withdrawn | 0 | 0 | 3
Not completed — Withdrawal by Subject | 53 | 51 | 55
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Study terminated by sponsor | 70 | 74 | 67
Not completed — Unavailability/noncompliance of study partner | 2 | 1 | 1
Not completed — Starting alternative treatment | 0 | 1 | 1
Not completed — Noncompliance with study procedures | 0 | 1 | 1
Not completed — Met stopping criteria | 0 | 0 | 1
Not completed — Health issues preventing continuation | 0 | 0 | 1
Not completed — Randomized in error, not treated | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were not collected from study partners.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo | Total
Number analyzed (Participants) | 376 | 374 | 375 | 1125
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.45 (7.624) | 73.64 (8.185) | 73.72 (7.926) | 73.94 (7.916)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 47 | 54 | 50 | 151
  65 to 74 years | 115 | 124 | 131 | 370
  ≥75 years | 214 | 196 | 194 | 604
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 208 | 214 | 629
  Male | 169 | 166 | 161 | 496
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 35 | 20 | 82
  Not Hispanic or Latino | 345 | 338 | 350 | 1033
  Unknown or Not Reported | 4 | 1 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 3 | 4
  Asian | 21 | 28 | 32 | 81
  Black or African American | 23 | 17 | 21 | 61
  White | 326 | 326 | 313 | 965
  Other | 1 | 1 | 4 | 6
  Multiple | 0 | 0 | 1 | 1
  Not reported | 4 | 1 | 1 | 6
  Unknown | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 46 | 47 | 56 | 149
  Puerto Rico | 6 | 9 | 4 | 19
  South Korea | 12 | 18 | 21 | 51
  United States | 312 | 300 | 294 | 906

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 12-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog12)
Description: The change from baseline to Week 76 in the ADAS-Cog12, a psychometrician-administered battery comprised of several cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Scores range from 0 (best) to 80 (worst).
Time Frame: Baseline (Study Day 1) to Week 76
Population: Data are from subjects in the modified intent-to-treat population (all randomized subjects with baseline plasma P-tau181 ≥44 pg/mL or other evidence of amyloid pathology, e.g., amyloid PET) who completed the assessment. No data were collected from study partners for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 167 | 181 | 188
score on a scale | 5.71 (0.529) | 5.65 (0.509) | 5.26 (0.506)
Statistical Analysis 1: Comparison: Simufilam 50 mg vs Placebo; Test type: Superiority; p = 0.5335, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.96 to 1.86]
Statistical Analysis 2: Comparison: Simufilam 100 mg vs Placebo; Test type: Superiority; p = 0.5836, Mixed Models Analysis; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.99 to 1.76]

2. Primary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL)
Description: The change from baseline to Week 76 in the ADCS-ADL, a 23-item study partner questionnaire that covers both basic activities of daily living (ADL) and more complex ADL or instrumental ADL for the subject. Scores range from 0 to 78, with a lower score indicating greater severity of functional loss.
Time Frame: Baseline (Study Day 1) to Week 76
Population: Data are from subjects in the modified intent-to-treat population (all randomized subjects with baseline plasma P-tau181 ≥44 pg/mL or other evidence of amyloid pathology, e.g., amyloid PET) whose study partner completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 169 | 179 | 187
score on a scale | -7.20 (0.646) | -6.87 (0.623) | -5.63 (0.620)
Statistical Analysis 1: Comparison: Simufilam 50 mg vs Placebo; Test type: Superiority; p = 0.0763, Mixed Models Analysis; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-3.30 to 0.17]
Statistical Analysis 2: Comparison: Simufilam 100 mg vs Placebo; Test type: Superiority; p = 0.1530, Mixed Models Analysis; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-2.93 to 0.46]

3. Secondary Outcome: Change From Baseline in the Integrated Alzheimer's Disease Rating Scale (iADRS)
Description: The change from baseline to Week 76 in the iADRS, where scores range from 0 to 146 with lower scores indicating worse performance.
Time Frame: Baseline (Study Day 1) to Week 76
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 167 | 177 | 185
score on a scale | -11.5 (0.901) | -11.5 (0.870) | -10.5 (0.865)

4. Secondary Outcome: Change From Baseline in the Neuropsychiatric Inventory (NPI)
Description: The change from baseline to Week 76 in the NPI, a 12-item study partner interview, which records the frequency and severity of common neuropsychiatric symptoms in dementia for the subject, as well as the level of study partner distress due to the neuropsychiatric problems. Scores range from 0 to 144, with higher scores indicating more frequent and severe symptoms, and greater levels of partner distress.
Time Frame: Baseline (Study Day 1) to Week 76
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 176 | 191 | 199
score on a scale | 1.57 (0.574) | 1.44 (0.556) | 0.37 (0.551)

5. Secondary Outcome: Change From Baseline in the MMSE
Description: The change from baseline to Week 76 in the MMSE, a set of standardized questions covering several target areas: orientation, registration, attention and calculation, short-term verbal recall, naming, repetition, 3-step command, reading, writing, and visuospatial cognitive assessment. Scores range from 0 to 30; lower scores indicate more severe impairment.
Time Frame: Baseline (Study Day 1) to Week 76
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 179 | 197 | 206
score on a scale | -3.48 (0.288) | -3.29 (0.277) | -3.35 (0.275)

6. Secondary Outcome: Change From Baseline in the Clinical Dementia Rating Sum of Boxes (CDR-SB)
Description: The change from baseline to Week 76 in the CDR-SB, which characterizes 6 domains of cognitive and functional performance applicable to AD and related dementias: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Scores for each domain have a minimum of 0 and a maximum of 3, and the 6 domain scores are summed to give the CDR-SB, which has a minimum score of 0 and a maximum score of 18. Higher scores indicate more severe impairment.
Time Frame: Baseline (Study Day 1) to Week 76
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 204 | 228 | 225
score on a scale | 1.65 (0.186) | 1.76 (0.187) | 1.84 (0.186)

7. Secondary Outcome: Change From Baseline in the Zarit Burden Interview (ZBI)
Description: The change from baseline to Week 76 in the ZBI, a 22-item study partner questionnaire designed to assess the stress or burden experienced by caregivers of people with dementia. Scores range from 0 to 88, with a higher score indicating greater stress or burden.
Time Frame: Baseline (Study Day 1) to Week 76
Population: Data are from the study partners of subjects in the modified intent-to-treat population (all randomized subjects with baseline plasma P-tau181 ≥44 pg/mL or other evidence of amyloid pathology, e.g., amyloid PET) who completed the assessment. No data were collected from study partners for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 169 | 180 | 185
score on a scale | 3.37 (0.734) | 4.68 (0.711) | 4.40 (0.706)

8. Other Pre Specified Outcome: Changes From Baseline in Brain Volume Via MRI
Description: Changes from baseline in hippocampus, ventricles, and whole brain volume.
Time Frame: Baseline (Study Day 1) to Week 76
Population: The overall number of subjects analyzed is the number of subjects who consented to take part in the MRI imaging substudy and for whom there was at least one non-missing post baseline MRI assessment available. MRIs were not conducted in the whole substudy population at Week 76. No data were collected from study partners for this outcome measure.
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 52 | 48 | 50
µL
  Whole brain volume | -17799.5 (13360.83) | -19043.6 (9721.20) | -17878.6 (14012.40)
  Ventricular volume | 5459.5 (4290.67) | 6109.9 (3766.34) | 6255.1 (5374.61)
  Hippocampal volume | -180.7 (109.82) | -192.2 (110.23) | -186.8 (114.54)

9. Other Pre Specified Outcome: Changes From Baseline in Amyloid Positron Emission Tomography (PET)
Description: Changes from baseline in amyloid deposition in the brain.
Time Frame: Baseline (Study Day 1) to Week 76
Population: The overall number of subjects analyzed is the number of subjects who consented to take part in the amyloid PET imaging substudy and for whom there were baseline and Week 76 values. No data were collected from study partners for this outcome measure.
Measure: Mean (Standard Deviation); unit: µL
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 31 | 19 | 27
µL | 0.0 (0.10) | 0.0 (0.09) | 0.0 (0.09)

10. Other Pre Specified Outcome: Changes From Baseline in Tau Positron Emission Tomography (PET)
Description: Changes from baseline in tau deposition in the brain
Time Frame: Baseline (Study Day 1) to Week 76
Population: The overall number of subjects analyzed is the number of subjects who consented to take part in the tau PET imaging substudy and for whom there were baseline and Week 76 values. No data were collected from study partners for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: µL
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 27 | 14 | 23
µL | 0.0 (0.10) | 0.0 (0.07) | 0.0 (0.10)

11. Other Pre Specified Outcome: Changes From Baseline in Plasma Biomarkers
Description: Change from baseline in the following plasma biomarkers of AD pathology, neurodegeneration, and neuroinflammation: phospho-tau217 (P-tau217), total tau, glial fibrillary acidic protein (GFAP), and neurofilament light chain (NfL).
Time Frame: Baseline (Study Day 1) to Week 76
Population: The overall number of subjects analyzed is the number of subjects who consented to take part in the plasma biomarker analysis substudy and for whom there were baseline and Week 76 values for each biomarker. Plasma samples were not obtained from the whole substudy population at Week 76. No data were collected from study partners for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 47 | 27 | 41
pg/mL
  Plasma P-Tau 217 | 43.6 (121.06) | 4.7 (15.74) | 4.0 (12.36)
  Plasma Total Tau | 50.7 (122.51) | 10.9 (41.92) | 7.0 (39.44)
  Plasma GFAP | 636.5 (1591.37) | 235.7 (846.47) | 107.7 (507.17)
  Plasma NfL | 872.3 (2023.12) | 321.3 (1397.74) | 351.4 (2075.46)

12. Other Pre Specified Outcome: Changes From Baseline in CSF Biomarkers
Description: Changes from baseline in CSF biomarkers of AD pathology, neurodegeneration, and neuroinflammation: P-tau217, total tau, GFAP, and NfL.
Time Frame: Baseline (Study Day 1) to Week 76
Population: The overall number of subjects analyzed is the number of subjects who consented to take part in the CSF biomarker analysis substudy and for whom there were baseline and Week 76 values for each biomarker. CSF samples were not obtained from the whole substudy population at Week 76. No data were collected from study partners for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 21 | 14 | 19
pg/mL
  CSF P-Tau 217 | 141.9 (169.08) | 90.5 (210.38) | 10.8 (139.20)
  CSF Total Tau | 136.7 (161.10) | 92.5 (152.32) | 28.7 (140.48)
  CSF GFAP | 1939.2 (2409.36) | 585.0 (2062.91) | 674.8 (1873.18)
  CSF NfL | 2372.6 (2494.67) | 1334.9 (2310.62) | 1535.9 (3383.45)

13. Other Pre Specified Outcome: Change From Baseline in Plasma Biomarker SavaDx
Description: Change from baseline in SavaDx, a novel plasma biomarker.
Time Frame: Baseline (Study Day 1) to Week 76
Population: Change from baseline in SavaDx, a novel plasma biomarker, was included in the protocol as part of the secondary analysis as a biomarker which may have been measured. The final SAP, which postdated the protocol, included the analysis of biomarkers as an exploratory/tertiary endpoint. However, analysis of SavaDx was not conducted due to a sponsor decision and therefore, no results are available.
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 78 weeks after subjects took their first dose of study drug, or until resolution or stabilization of any AEs ongoing at the end of the study.
Description: Data are from the safety population, which included all subjects who received at least 1 dose of study drug. Study partners were not part of the safety population. No AE data were collected from study partners.
Arm/Group | Simufilam 50 mg | Simufilam 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 6/376 | 2/374 | 3/373
Serious Adverse Events (participants affected / at risk) | 61/376 | 43/374 | 45/373
Other Adverse Events (participants affected / at risk) | 198/376 | 184/374 | 195/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simufilam 50 mg (N=376) | Simufilam 100 mg (N=374) | Placebo (N=373)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 1 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simufilam 50 mg (N=376) | Simufilam 100 mg (N=374) | Placebo (N=373)
COVID-19 (Infections and infestations) | 47 (48) | 43 (43) | 38 (38)
Urinary tract infection (Infections and infestations) | 39 (47) | 32 (40) | 34 (43)
Nasopharyngitis (Infections and infestations) | 7 (8) | 10 (11) | 9 (12)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 6 (6) | 6 (8)
Dizziness (Nervous system disorders) | 11 (11) | 26 (29) | 22 (25)
Headache (Nervous system disorders) | 16 (22) | 17 (18) | 13 (15)
Syncope (Nervous system disorders) | 4 (4) | 0 (0) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 19 (19) | 14 (18) | 15 (17)
Nausea (Gastrointestinal disorders) | 9 (9) | 13 (19) | 15 (15)
Constipation (Gastrointestinal disorders) | 6 (7) | 11 (11) | 11 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 4 (4) | 7 (7)
Vomiting (Gastrointestinal disorders) | 5 (5) | 8 (12) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 40 (56) | 32 (50) | 48 (64)
Contusion (Injury, poisoning and procedural complications) | 8 (8) | 6 (7) | 5 (5)
Anxiety (Psychiatric disorders) | 14 (14) | 13 (13) | 12 (13)
Depression (Psychiatric disorders) | 12 (12) | 9 (9) | 16 (16)
Agitation (Psychiatric disorders) | 16 (16) | 5 (7) | 14 (15)
Insomnia (Psychiatric disorders) | 8 (8) | 8 (8) | 6 (6)
Confusional state (Psychiatric disorders) | 6 (6) | 8 (8) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 12 (12) | 13 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 13 (13) | 9 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2) | 3 (3)
Weight decreased (Investigations) | 6 (6) | 17 (18) | 8 (8)
Fatigue (General disorders) | 15 (15) | 16 (16) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 8 (8) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (10) | 7 (10)
Hypertension (Vascular disorders) | 11 (11) | 5 (5) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and PI must request review and comment of any proposed publication by the sponsor at least 90 days prior to submission of the publication. The sponsor will advise of any information which is confidential information or which may impair the sponsor's ability to obtain patent protection, and has the right to require confidential information or factual errors to be removed, or to delay the proposed publication by an additional 90 days to allow the sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT05026177/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT05026177/SAP_001.pdf